CLINICAL TRIAL: NCT00276146
Title: Dipyridamole/Magnesium To Improve Sickle Cell Hydration
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The NHLBI BSMB recommended closure due to poor enrollment.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: CCHMC 03-7-41; U54HL070871 (NIH)
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Anemia, Sickle Cell
Keywords: dipyridamole; magnesium; sickle cell; anemia; red blood cells
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia | interventions — Dipyridamole; Magnesium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: oral dipyridamole, oral magnesium, or a combination of both

SUMMARY:
The purpose of this study is to determine the benefits as well as side effects of giving drugs called dipyridamole and magnesium to patients with sickle cell anemia (SCA).

DETAILED DESCRIPTION:
Vaso-occlusive episodes are the most common problem experienced by patients with SCA and the most frequent reason for hospital admissions as well as visits to the clinic and emergency department. Many cellular, humoral, and vascular factors influence the initiation and propagation of vaso-occlusion by sickle cells. Among these is the tendency of sickle cells (SS RBC) to become dehydrated with accompanying increase in the hemoglobin (Hb) concentration. Since sickle hemoglobin (Hb S) concentration controls the rate of polymerization, cellular dehydration plays a key role in sickle cell pathology.

Two separate but interdependent cation transport mechanisms affect sickle cell hydration, the first involving abnormal KCl cotransport (KCC), and the second a sickle-induced (SI) passive leak which permits the influx of calcium ions (Ca++) that activates the Gardos pathway, a Ca++-dependent K channel. Early investigations aimed at inhibiting KCC with magnesium (Mg) and the Gardos pathway with clotrimazole met with partial success. We have recently shown in vitro that dipyridamole also inhibits the SI pathway. Strategies designed to block the formation of these dense, dehydrated cells would offer important therapeutic options that might decrease the number and severity of the vaso-occlusive episodes in patients. Drawing on the information gained from two decades of research on cation transport in SS RBC, including the unique discovery made at this Center that dipyridamole inhibits the SI cation leak, we now propose a study of combined therapy using two transport inhibitors aimed at reducing SS RBC dehydration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with homozygous sickle cell (Hb SS) confirmed by hemoglobin electrophoresis or HPLC
* Patients with adequate cardiac, renal, and liver function
* Patients with baseline fetal hemoglobin (Hb F) level of 10% or less
* Patients with at least 6% dense cells or higher at initial screening visit
* Patients with no history of coronary heart disease
* Patients with normal baseline ECG
* Patients with no history of hypotension or hypotensive episodes

Exclusion Criteria:

* Patients who are pregnant, trying to become pregnant, or breast feeding
* Patients who are on a chronic transfusion program
* Patients who are unable to take oral medications
* Patients who have significant cardiac, renal, or liver dysfunction
* Patients who are on hydroxyurea
* Patients who have a fetal hemoglobin (Hgb F) level of greater than 10%, or have less than 6% dense cell on initial screen
* Patients who are taking a supplement which contains magnesium
* Patients who are taking aspirin, ibuprofen on a daily basis, or anti-coagulant such as Coumadin on a daily basis
* Patients who have a known underlying coagulopathy (acquired or congenital) or have prolonged PT or PTT at the time of initial screen
* Patients who have had a hypersensitivity to either of the study medications
* Patients who are taking any other study medication(s). Patients will not be excluded if they are on penicillin prophylaxis or folic acid, or use ibuprofen intermittently
* Patients taking tetracycline or sodium polystyrene sulfonate
* Patients on concomitant medications and other therapy must have a wash out period prior to study entry and/or study drug dosing
* Patients with abnormal baseline ECG
* Patients with a history of hypotension or hypotensive episodes

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-05

PRIMARY OUTCOMES:
To assess effects on red cell hydration.
To assess effects on red cell survival. Measurements will be performed before and after treatment.

SECONDARY OUTCOMES:
To monitor side effects of each treatment arm.
To evaluate clinical outcomes during each phase of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Kalinyak, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Cincinnati, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

REFERENCES:
- See also: Sickle Cell Center at Cincinnati Children's Hospital Medical Center — http://www.cincinnatichildrens.org/svc/alpha/b/blood/programs/sickle-cell/